CLINICAL TRIAL: NCT05840640
Title: Granulocyte Colony Stimulating Factor Four Week Plus N-Acetyl Cysteine in Severe Alcoholic Hepatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Former Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCSF IN SAH
Record Dates: First submitted 2023-04-17; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Alcoholic Hepatitis
Keywords: alcoholic hepatitis; alcoholic liver disease; regeneration
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Diseases, Alcoholic | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: Open label randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Medical therapy (Active Comparator): Standard medical therapy involves primary treatment with normal hospital nutrition (1800 to 2000 kcal per day). Diuretics, sodium restriction and albumin for treatment of ascites or fresh frozen plasma for coagulopathy or antibiotics for any focus of infection as spontaneous bacterial peritonitis (SBP), pneumonia, cellulitis, and urinary tract infection as indicated.
  Interventions: Drug: Standard Medical Therapy
- G-CSF (Experimental): Standard Medical Therapy plus G-CSF- 5μg/Kg s.c every 12 hours for 5 consecutive days
  Interventions: Drug: Standard Medical Therapy; Drug: G-CSF
- G-CSF and NAC (Experimental): Standard Medical Therapy plus G-CSF with intravenous NAC (day 1: NAC at 150, 50, and 100 mg/kg in 250, 500, and 1000 ml of 5% glucose solution over 30 minutes, 4 hours, and 16 hours, respectively; days 2 through 5: 100 mg/kg/day in 1000 ml of 5% glucose solution followed by oral NAC from days 6 to 28)
  Interventions: Drug: Standard Medical Therapy; Drug: G-CSF; Drug: G-CSF and NAC

INTERVENTIONS:
Drug: Standard Medical Therapy — Standard medical therapy involves primary treatment with normal hospital nutrition (1800 to 2000 kcal per day). Diuretics, sodium restriction and albumin for treatment of ascites or fresh frozen plasma for coagulopathy or antibiotics for any focus of infection as spontaneous bacterial peritonitis (SBP), pneumonia, cellulitis, and urinary tract infection as indicated.
Drug: G-CSF — standard medical therapy plus G-CSF- 5μg/Kg s.c every 12 hours for 5 consecutive days
  Arms: G-CSF; G-CSF and NAC
Drug: G-CSF and NAC — Standard Medical Therapy plus G-CSF with intravenous NAC (day 1: NAC at 150, 50, and 100 mg/kg in 250, 500, and 1000 ml of 5% glucose solution over 30 minutes, 4 hours, and 16 hours, respectively; days 2 through 5: 100 mg/kg/day in 1000 ml of 5% glucose solution followed by oral NAC from days 6 to 28)
  Arms: G-CSF and NAC

SUMMARY:
Alcoholic hepatitis is related to very high mortality rate. About 40% of the patients died within first 6 months after the detection of the clinical syndrome. Therefore, it is very essential for proper diagnosis and early treatment . In response to acute or chronic liver damage, bone marrow derived stem cells can spontaneously populate liver and differentiate into hepatic cells. Animal and human studies suggested that injured hepatocyte may be replaced by pluripotent bone marrow cells. However, this hepatocyte repopulation is highly dependent on varieties of liver injury and therapeutic conditions. The studies have suggested Granulocyte-colony stimulating factors (G-CSF) can regenerate hepatocyte by fusing with hematopoietic cells, thereby enhancing the liver histology and survival rate.

G-CSF is a cytokine capable to regulate a number of functions in neutrophils. In three recent studies mobilization of bone marrow stem cells induced by G-CSF was observed in patients with alcoholic hepatitis. In two of these studies there was a survival benefit with the use of G-CSF.

Alcoholism leads to decrease in endogenous antioxidant potential. Alcoholic liver disease (ALD) patients show low endogenous antioxidants. Chronic ethanol consumption cause selective deficiency in the availability of reduced glutathione (GSH) in mitochondria has been reported. This is due to impaired functioning of GSH transporter from cytosol to mitochondrial matrix. The effect on glutathione replenishing potential by N-acetyl cysteine (NAC) can be used to reduce oxidative stress, which also has excellent safety profile. Therefore, NAC can be used for severe alcoholic hepatitis treatment due to its therapeutic potential factor. NAC also inhibit apoptosis and pro-inflammatory cytokine production. In a study high doses of intravenous N-acetyl cysteine therapy for 14 days conferred neither survival benefits nor early biological improvement in severe acute alcoholic hepatitis patients with adequate nutritional support.However, these results must be viewed with caution, since the study suffered from a lack of power. In a recent study, NAC and corticosteroids combination therapy benefits among patients with severe acute alcoholic hepatitis in 1 month survival, although the final outcome at 6 month survival was not improved. There are no studies on the use of combination therapy of 4 weeks of NAC plus G-CSF in patient with severe alcoholic hepatitis.

Therefore the investigators plan to study the safety and efficacy of combination therapy of G-CSF and 4 weeks of NAC in the patients with alcoholic hepatitis.

ELIGIBILITY:
Inclusion Criteria:

• Alcoholic hepatitis patients(More than 10 years of heavy alcohol consumption (mean intake ≈ 100 g/day);Elevated aspartate aminotransferase level (but <500 IU per millilitre) and Ratio ofAST/ALT≥2 times;Elevated serum total bilirubin level ≥ 5 mgdL (86 μmol/L);Elevated INR(≥1.5) and;Neutrophilia. Patient with Maddrey's DF of≥ 32 will be included in the study, with or without biopsy)

Exclusion Criteria:

* Age < 18 and > 75 years
* Hepatocellular carcinoma or portal vein thrombosis
* Refusal to participate in the study
* Serum creatinine >1.0 mg%
* Hepatic encephalopathy- grade 3 or 4
* Upper gastrointestinal bleed in last ten days
* Uncontrolled bacterial infection
* Human immunodeficiency virus, Hepatitis B virus, Hepatitis C virus seropositivity, Autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha1-antitrypsin deficiency
* Pregnancy
* Glucocorticoid treatment
* Significant co-morbidity
* Previous known hypersensitivity to G-CSF/NAC

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Survival at the end of 90 days | 90 days

SECONDARY OUTCOMES:
Number of CD34+ cells in peripheral blood | 6 days
Change in MELD score | 90 days
Change in modified Maddrey's Discriminant Function at 90 days. | 90 days
  Modified Maddrey's Discriminant Function will be calculated using the following formula:
  [4.6 × (prothrombin time of patient - prothrombin time of control) + serum bilirubin in mg/dl]
  Modified Maddrey's Discriminant Function is a validated and well-established parameter for assessing the severity and prognosis of alcoholic hepatitis.
Change in Child Turcotte Pugh score | 90 days
Number of participants with treatment-related adverse events in the different treatment groups | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Hepatology, PGIMER, Chandigarh, India